CLINICAL TRIAL: NCT07380438
Title: A Clinical Study to Evaluate the Efficacy of Nutritional Supplements on Human Health and to Assess the Reliability of Sponsor's Device
Brief Title: A Clinical Study to Evaluate the Efficacy of a Nutritional Supplement to Improve Carotenoid Content as Measured by a Non-invasive Hyperspectral Absorption Device
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pharmanex (Industry)
Collaborators: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 25-K540049EPE
Record Dates: First submitted 2026-01-04; First posted 2026-02-02 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2026-01

CONDITIONS: Nutrition Assessment
Keywords: antioxidant; carotenoid

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active (Active Comparator): LifePak Optimum nutritional supplement
  Interventions: Dietary Supplement: LifePak Optimum nutritional supplement
- Placebo (Placebo Comparator): Placebo supplement
  Interventions: Dietary Supplement: Placebo supplement

INTERVENTIONS:
Dietary Supplement: LifePak Optimum nutritional supplement — Ca(mg) Vit C(mg) Mg(mg) Se(㎍) Cr(㎍) Vit E(mg a-TE) Mo(㎍) Pantothenic acid(mg) Vit B12(㎍) Niacin(mgNE) Zn(mg) Vit B6(mg) Biotin(㎍) Vit D(㎍) Vit B1(mg) Vit B2(mg) Cu(mg) Mn(mg) Vit K(㎍) Folic acid(㎍)_Folic acid Iodine(㎍) Beta-carotene(mg) Lycopene(mg) Lutein(mg)
  Arms: Active
Dietary Supplement: Placebo supplement — Placebo supplement
  Arms: Placebo

SUMMARY:
The goal of this clinical trial is to evaluate a nutritional supplement in an otherwise healthy adult population. The main questions it aims to answer are:

* Do antioxidant carotenoid levels increase in after supplementation as measured by a non-invasive device?
* Do wellness factors correlate with supplementation?

Researchers will compare the nutritional supplement arm to a placebo group to assess its effects.

Participants will take either the nutritional supplement or placebo once daily for 8 weeks. Participants will be scanned by a non-invasive hyperspectral absorption device to obtain a skin carotenoid score. Participants will also have facial images taken, dermal spectrophotometry measurements of their face, and complete self-assessment questionnaires.

ELIGIBILITY:
Inclusion Criteria:

* Aged 20-60 years.
* all skin types
* BMI between 18.5-23
* No allergy with carotenoid-containing supplements

Exclusion Criteria:

* subject who have undergone organ excision, organ transplantation, or experienced a skull concussion with extended loss of consciousness in the past 5 years, or with current after effects.
* subjects with diseases such as heart disease, myocardial infarction, cancer, tuberculosis, chronic or acute renal failure, poliomyelitis, arthritis, or asthma
* Subjects undergoing or schedule for long-term treatment, particularly with anti-inflammatory agents, steroids, sedatives, diabetes treatments, medications for blood pressure, hormone therapies, antihistamines, and/or drugs with similar functions,
* subjects who have taken contraceptives or herbal medicines continuously for more than 2 months within the past 3 weeks,
* subjects with any current medical condition, including gynecological disorders, or those undergoing hospital treatment,
* subjects with known allergies to aspirin, antibiotics, fruits, laboratory substances, sunlight or metals;
* Subjects who experience herpes outbreaks more than five times a year or suffer from acute swelling of the skin or mucous membranes;
* Subjects with a history of psychiatric disorders, including sleep disorders or panic disorder

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 84 (Actual)
Dates: Start 2025-10-20 (Actual); Primary Completion 2025-11-20 (Actual); Study Completion 2026-01-08 (Actual)

PRIMARY OUTCOMES:
Skin carotenoid score via Prysm iO device | 8 weeks
  The Prysm iO device will provide a numerical score between 0-1000. The score is an indicator of skin carotenoid concentration/nutritional wellness. The higher the score the more positive the outcome.
Short-Form 36 Health Survey | 8 weeks
  The Short-Form 36 Health Survey is a validated questionnaire that measures multidimensional health-related quality of life, including specific domains of everyday life. The questionnaire has a 1-5 scale, with the higher score reflected a better perception of health-related outcomes.
Skin color measurement via Spectrophotometer | 8 weeks
Perceived Immunity | 8 weeks
  Perceived Immunity Scale, a validated questionnaire to assess individuals' beliefs about the strength of their immune system. The assessment uses a 1-6 point Likert scale, where a lower score indicates greater disagreement with the statement, and a higher score indicates greater agreement with the statement.
Psychological Scales Related to Physical Condition | 8 weeks
  Short Health Anxiety Inventory (SHAI) a validated questionnaires using a 1-5 point Likert scale, (where a lower score indicates greater disagreement, and higher score indicates greater agreement) to assess feelings about health and recovery.
Fatigue and Vitality Status Assessment | 8 weeks
  Multi-Dimensional Fatigue Inventory--a validated questionnaire using a 1-7 Likert scale (where a lower score indicates greater disagreement, and a higher score indicates greater agreement) to assess an individual's fatigue state.
Brief Resilience Scale (BRS) | 8 weeks
  The Brief Resilience Scale (BRS) is a validated questionnaire, using a 1-5 point Likert scale (where a lower score indicates greater disagreement, and a higher score indicates greater agreement), to assess the ability to bounce back from feelings of stress.

CONTACTS AND LOCATIONS:
Locations (1):
- I.E.C. Korea, Suwon, Gyeonggi-do, South Korea

IPD SHARING:
Plan to Share IPD: Undecided